CLINICAL TRIAL: NCT05749666
Title: A Prospective Randomized Double-blinded Controlled Single Center Clinical Study of the Efficacy and Safety for Tofacitinib Compared With Glucocorticoid in the Remission-reduction Treatment of Active Takayasu's Arteritis
Brief Title: Comparison of Tofacitinib and Prednisolone in the Treatment of Active Takayasu's Arteritis
Acronym: TOFGCTAK
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Principal Investigator, Xinping Tian, Professor of Medicine, Chinese SLE Treatment And Research Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSTAR-009
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Takayasu Arteritis
Keywords: Tofacitinib; prednisolone
MeSH Terms: conditions — Takayasu Arteritis | interventions — tofacitinib; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tofacitinib group (Experimental): Tofacitinib 5mg BID taken orally for 24 weeks and placebo of prednisolone taken daily according to preset tapering protocol during same period
  Interventions: Drug: Tofacitinib 5 MG; Other: Placebo of prednisolone
- Prednisolone group (Active Comparator): Prednisolone taken daily according to preset tapering protocol and placebo of tofacitinib 5mg BID taken orally for 24 weeks
  Interventions: Drug: Prednisolone; Other: Placebo of tofacitinib 5mg

INTERVENTIONS:
Drug: Tofacitinib 5 MG — Tofacitinib 5 MG BID taken orally for 24 weeks
  Arms: Tofacitinib group
Drug: Prednisolone — Prednisolone taken daily according to preset tapering protocol
  Arms: Prednisolone group
Other: Placebo of tofacitinib 5mg — Placebo of tofacitinib 5mg BID taken orally for 24 weeks
  Arms: Prednisolone group
Other: Placebo of prednisolone — Placebo of prednisolone taken daily according to preset tapering protocol for 24 weeks
  Arms: Tofacitinib group

SUMMARY:
This is a prospective, double-blinded, single center, randomized clinical trial. It compares the clinical efficacy and safety of thees 2 drugs in the treatment of active Takayasu's arteritis patients.

DETAILED DESCRIPTION:
In this study, 40 Takayasu's arteritis patients with active disease will be enrolled. Patients are randomized into the tofacitinib treatment group and prednisolone treatment group. Patients will follow the same reduction steps for prednisolone and its placebo. The primary end point is the percentage of patients who are in complete response at week 24.

The efficacy will be evaluated at week 4, 12 and 24. Safety is also monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18-65 years old;
2. Fulfilled the classification criteria of Takayasu's arteritis by ACR 1990;
3. Active TAK: defined by the definition of active disease in the recommendations released by EULAR in 2018 or Kerr's criteria by NIH;
4. Patients who signed the informed consent form.

Exclusion Criteria:

1. Patients who failed or intolerant to either tofacitinib or its similar drugs;
2. Patients with severe liver disease defined by the serum ALT or AST elevated more than 2 times the upper limits;
3. Not well controlled diabetes;
4. Moderate and severe hyperlipedimia;
5. Patients with history of thrombus;
6. Uncontrolled heart failure od renal dysfunction (eGFR <30ml/min);
7. Patients with active infection, including tuberculosis, hepatitis B and C, HIV infection, bacterial or fungal infection;
8. Upper GI bleeding happened in 3 months before enrollment;
9. Refractory hypertension;
10. Pregnant or intended to be pregnant recently;
11. Severe coronary artery involvement demonstrated by CTA;
12. Severe cranial or cervical or renal artery diseases that need surgery;
13. Patients that should not be included judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete response | week 24
  Percentage of patients with complete response at week 24

SECONDARY OUTCOMES:
Percentage of patients with partial response | week 24
  Percentage of patients with partial response at week 24
Percentage of patients with adverse events due to treatment of tofacitinib | 24 weeks
  Percentage of patients with adverse events due to treatment of tofacitinib at week 24
Percentage of patients with adverse events due to treatment of prednisolone | 24 weeks
  Percentage of patients with adverse events due to treatment of prednisolone at week 24
Percentage of patients with progression, no change, and improvement in vessel image at the end of study | week 24
  Percentage of patients with progress disease, stable disease, and improved disease demonstrated by CTA, MRI or Doppler at week 24
Intervention procedures | 24 weeks
  Percentage of patients who require intervention procedures during the study period
Complication of Takayasu's arteritis | 24 weeks
  Complication of Takayasu's arteritis happened during 24 weeks
Glucocorticoid toxicity index | week 24
  Glucocorticoid toxicity index at week 24 which indicate the toxicity of prednisolone.

CONTACTS AND LOCATIONS:
Overall Officials: Xinping Tian, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China